CLINICAL TRIAL: NCT05156541
Title: Open Controlled Randomized Study of the Efficacy and Safety of Ingaron (Interferon-gamma) in the Treatment of Anogenital Warts (Phase III)
Brief Title: Study of the Efficacy and Safety of the Drug Ingaron (Interferon-gamma) in the Treatment of Anogenital Warts
Acronym: ING-HPV-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SPP Pharmaclon Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ING-HPV-1
Record Dates: First submitted 2021-11-15; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Human Papillomavirus Infection; Anogenital Warts
Keywords: interferon gamma; IFN-g; HPV; Anogenital warts
MeSH Terms: conditions — Papillomavirus Infections; Condylomata Acuminata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interferon (Experimental): After a cryodestruction session, therapy with Ingaron 100,000 IU once a day every other day. The course of treatment consisted of 5 injections.
  Interventions: Drug: Interferon gamma human recombinant (IFN-G)
- Control (No Intervention): Cryodestruction session only.

INTERVENTIONS:
Drug: Interferon gamma human recombinant (IFN-G) — received by microbiological synthesis; specific antiviral activity on cells is 2x10*7 Units per mg of protein
  Other Names: Ingaron; Interferon gamma human recombinant
  Arms: Interferon

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness of destructive therapy for anogenital warts in combination with the use of Ingaron in comparison with destructive therapy.

DETAILED DESCRIPTION:
Literature data and the results of preclinical studies of interferon-gamma, as well as the features of HPV immunopathogenesis, show the expediency of studying the use of Ingaron in this pathology.

The study was planned to include 50 outpatients of both sexes aged 18 to 50 years with a confirmed diagnosis of anogenital warts.

In the course of the study, Ingaron was administered at a dose of 100,000 IU once a day every other day in the period of 10 days.

Patients were divided into 2 groups: study and control.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged 18 to 50 years with a diagnosis of "Anogenital warts".
2. The diagnosis "Anogenital warts" was made for the first time at least one year before inclusion in the study.
3. During the last year prior to inclusion in the study, the patient had at least 2 recurrences of anogenital warts.
4. The diagnosis is confirmed by the detection of HPV by polymerase chain reaction (PCR).
5. Negative pregnancy test in women.
6. Availability of written informed consent to participate in the study.

Exclusion Criteria:

1. Positive test results for syphilis, hepatitis (HbsAg, anti-HCV), HIV infection, gonococcal infection, urogenital trichomoniasis, chlamydial infection, inflammatory diseases of the urogenital system caused by genital mycoplasmas.
2. Unsystematic use of barrier methods of contraception.
3. Pregnancy and lactation.
4. Known allergic reactions to interferons and / or other significant allergic diseases.
5. Any immunotropic therapy within the last 6 weeks prior to enrollment in the study.
6. The need to take drugs prohibited during the study.
7. Condition after organ transplantation, constant intake of immunosuppressive drugs.
8. Severe pathology from the cardiovascular system (uncontrolled arterial hypertension, unstable angina pectoris, congestive heart failure, cardiac arrhythmias), a history of myocardial infarction or cerebrovascular accident within the last 6 months.
9. Severe pathology on the part of the liver (increased content of AST, ALT 2 times higher than the upper limit of the norm, the content of total bilirubin> 2 mg / dL), kidney (content of creatinine> 1.5 mg / dL); signs of hepatic and / or renal failure.
10. The presence of severe pathology on the part of the respiratory system, gastrointestinal tract, hematopoietic system.
11. Other serious (acute or chronic) pathological conditions, including mental illness, as well as abnormalities in laboratory parameters, which, in the opinion of the investigator, may increase the risk associated with participation in the study or affect the interpretation of efficacy and safety data obtained in this research.
12. Alcohol and / or drug dependence.
13. Participation in other clinical trials in the last three months prior to inclusion.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05-18 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2010-07-15 (Actual)

PRIMARY OUTCOMES:
Recurrence of anogenital warts | Day 11
  Number of participants with recurrent anogenital warts
Recurrence of anogenital warts | Day 40
  Number of participants with recurrent anogenital warts
Recurrence of anogenital warts | Day 100
  Number of participants with recurrent anogenital warts

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Apanansky, Master, Study Director — SPP Pharmaclon Ltd.
Locations (1):
- State scientific center of a dermatovenereology and cosmetology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No